CLINICAL TRIAL: NCT00460577
Title: Randomized, Double Blind, Double Dummy, Placebo Controlled Trial to Compare the Effectiveness of Formoterol vs Ipatropioum Bromide Plus Fenoterol in Asthmatic Children (5-<12 Years) With Acute Bronchial Obstruction Attending Emergency Services
Brief Title: Efficacy of Formoterol vs Ipatropioum Bromide Plus Fenoterol in Children (5-<12 Years) With Acute Bronchial Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CFOR258DVE02
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Acute Bronchial Obstruction, Asthma
Keywords: Asthma, Formoterol, Bronchial Obstruction, Children
MeSH Terms: conditions — Asthma | interventions — Fenoterol; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Formoterol (Foradil®) (Active Comparator): Formoterol (Foradil®) 12 micrograms administered through Aerolizer®.
  Interventions: Drug: Formoterol fumerate
- Fenoterol 0.5 mg + Ipratropium Bromide (Berodual®) 0.25 mg (Active Comparator): Fenoterol 0.5 mg + Ipratropium Bromide (Berodual®) 0.25 mg 20 drops in 3 mL of saline solution nebulized.
  Interventions: Drug: fenoterol/ipratropium bromide

INTERVENTIONS:
Drug: Formoterol fumerate — 12 micrograms stat (twice if necessary). Inhaled via aerolizer
  Arms: Formoterol (Foradil®)
Drug: fenoterol/ipratropium bromide — 0.5 micrograms/0.25 milligrams (20 drops) inhaled via nebulization diluted in 3cc of 0.9% saline.
  Arms: Fenoterol 0.5 mg + Ipratropium Bromide (Berodual®) 0.25 mg

SUMMARY:
To determine efficacy and tolerability of inhaled Formoterol vs nebulized Ipatropioum Bromide plus Fenoterol in cumulative sequential doses in asthmatic children (5-<12 years) with acute bronchial obstruction attending emergency services

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic children 5-<12 years old, requiring emergency services for acute bronchial obstruction mild to moderate determined by functional and clinical evidence

Exclusion Criteria:

* Patients with severe acute bronchial obstruction determined by functional and clinical evidence
* Patients unable to use the inhaling device at time of treatment
* Patients who received a bronchodilator drug within the last 12 hours
* Patients who received inhaled steroids within the last 72 hours
* Patients who received systemic steroids within the last 7 days
* Patients with near fatal asthma history
* Patients with fever (>38.5°C axillar temp)
* Patients with any clinical significance condition

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis de Venezuela, Study Chair — Novartis de Venezuela
Locations (2):
- Venezuela (2):
  - Novartis Investigator site - five sites in Caracas, Caracas
  - Novartis Investigator Site, Maracaibo

RESULTS

PARTICIPANT FLOW:
Groups:
- Fenoterol 0.5 mg + Berodual®: Fenoterol 0.5 mg + Ipratropium Bromide (Berodual®) 0.25 mg 20 drops in 3 mL of saline solution nebulized.
Period: Overall Study
Arm/Group | Formoterol (Foradil®) | Fenoterol 0.5 mg + Berodual®
Started | 30 (148 patients were screened; however, 22 did not consent and 66 did not meet inclusion/exclusion.) | 30
Completed | 28 | 24
Not Completed | 2 | 6
Not completed — Protocol Violation | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Formoterol (Foradil®) | Fenoterol 0.5 mg + Berodual® | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.8 (1.5) | 7.8 (2.1) | 7.8 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 18 | 19 | 37
Maximum Inspiratory Flow [Mean (Standard Deviation); unit: Liters/minute] — Mean of the Maximum Inspiratory Flow
  Liters/minute | 77.7 (16.7) | 79.9 (17.5) | 78.8 (0)
Maximum Expiratory Flow [Mean (Standard Deviation); unit: Liters/minute] — Mean of Maximum Expiratory Flow
  Liters/minute | 140.3 (33.1) | 150.3 (36.6) | 145.3 (0)
Forced Expiratory Flow 1 sec [Mean (Standard Deviation); unit: Liters] — Mean of Forced Expiratory Flow one second (FEV1) defined as the volume of air that can be forced out in 1 second after taking a deep breath.
  Liters | 1.06 (0.280) | 1.12 (0.289) | 1.09 (0)
Forced Expiratory Flow 1 sec as a Percentage of Predicted [Mean (Standard Deviation); unit: Percentage of Predicted] — Mean Expiratory Flow 1 second as a Percentage of Predicted
  Percentage of Predicted | 67.05 (15.22) | 71.17 (15.76) | 69.11 (0)
Conway Clinical Scale [Mean (Standard Deviation); unit: score on a scale] — Mean of Clinical Scale score measured by assessment of the following: Wheezing, Accessory Muscle Use and Pulse Frequency in a 0 to 3 point scale according to severity for a minimum of 0 points and a total of 9 points in a very severe clinical case.
  score on a scale | 4.1 (1.4) | 4.0 (1.5) | 4.05 (0)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Maximum Expiratory Flow From Baseline to Final Evaluation
Description: Mean Change from Baseline to Final Evaluation in the Per Protocol population assessed by Maximum Expiratory Flow.
Time Frame: Baseline,4 hours
Population: Per protocol population: defined as number of patients who did not present any major deviations from protocol and received at least one dose of investigational study drug.
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Formoterol (Foradil®) | Fenoterol 0.5 mg + Berodual®
Number analyzed (Participants) | 28 | 24
Liters/minute | 44 (26.87) | 43.67 (20.48)

2. Secondary Outcome: Safety Assessed by: Pulse Oxymetry, Clinical Assessments, Adverse Events
Description: Not posted: see comment in Limitations and Caveats.
Time Frame: 4 hours
Reporting Status: Not Posted
Measure: Number; unit: Participants

3. Secondary Outcome: Pharmacoeconomic Analysis
Description: Pharmacoeconomic analysis comparing the mean direct costs (total cost per prescription) of treatment with Formoterol (Foradil®) to treatment with Fenoterol 0.5 mg + Berodual®.
Time Frame: 4 hours
Population: as for outcome 1
Measure: Mean (Full Range); unit: Cost in US Dollars
Arm/Group | Formoterol (Foradil®) | Fenoterol 0.5 mg + Berodual®
Number analyzed (Participants) | 28 | 24
Cost in US Dollars | 9.21 [6.19 to 12.93] | 25.67 [21.95 to 29.91]

4. Primary Outcome: Mean Change in Forced Expiratory Volume in 1 Second (FEV1) From Baseline to Final Evaluation
Description: Mean Change from Baseline to Final Evaluation in the Per Protocol population assessed by Forced Expiratory Volume in 1 second. FEV1 is defined as the volume of air that can be forced out of the lungs in 1 second after taking a deep breath.
Time Frame: Baseline,4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Formoterol (Foradil®) | Fenoterol 0.5 mg + Berodual®
Number analyzed (Participants) | 28 | 24
Liters | 0.32 (0.2) | 0.34 (0.22)

5. Primary Outcome: Mean Change in Pulse Oxymetry From Baseline to Final Evaluation
Description: Mean Change from Baseline to Final Evaluation in the Per Protocol population assessed by Pulse Oximetry used to monitor the percentage of oxygen saturation of hemoglobin in the blood.
Time Frame: Baseline, 4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Formoterol (Foradil®) | Fenoterol 0.5 mg + Berodual®
Number analyzed (Participants) | 28 | 24
percentage | 2.57 (1.67) | 2.83 (2.51)

6. Primary Outcome: Mean Change in the Conway Clinical Scale Score From Baseline to Final Evaluation
Description: Mean Change from Baseline to Final Evaluation in the Per Protocol population assessed by the Conway Clinical Scale. Assessment of the following: Wheezing, Accessory Muscle Use and Pulse Frequency in a 0 to 3 point scale according to severity for a minimum of 0 points and a total of 9 points in a very severe clinical case.
Time Frame: Baseline,4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Formoterol (Foradil®) | Fenoterol 0.5 mg + Berodual®
Number analyzed (Participants) | 28 | 24
score on a scale | -3.18 (1.59) | -3.04 (1.83)

ADVERSE EVENTS:
Arm/Group | Formoterol (Foradil®) | Fenoterol 0.5 mg + Berodual®
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Secondary Outcome Measure 2: Safety Assessed by Pulse Oxymetry, Clinical Assessments, Adverse Events has not been posted. Analysis of Pulse Oxymetry and Clinical Assessment was not performed. Adverse events are reported in the Adverse Event section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.